CLINICAL TRIAL: NCT00111566
Title: Brief Infusion of Eptifibatide Following Percutaneous Coronary Intervention
Brief Title: BRIEF-PCI: Brief Infusion of Eptifibatide Following Percutaneous Coronary Intervention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cardiology Research UBC (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, Anthony Fung, MD, Principal Investigator, Cardiology Research UBC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C04-0359
Record Dates: First submitted 2005-05-23; First posted 2005-05-24 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
Keywords: Percutaneous Coronary Intervention (PCI); Glycoprotein IIb/IIIa blockade; Ischemic complications following PCI
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction | interventions — Eptifibatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 18 Hour infusion (Active Comparator)
  Interventions: Drug: eptifibatide
- 4 hour infusion (Experimental)
  Interventions: Drug: eptifibatide

INTERVENTIONS:
Drug: eptifibatide

SUMMARY:
This trial was designed to examine the efficacy of a brief versus a standard prolonged (18 hours) infusion of eptifibatide in preventing troponin I release following successful coronary stenting.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) is a common treatment for patients with severe ischemic heart disease. In the majority of cases, the potent anti-platelet agent eptifibatide is administered (bolus followed by infusion for 18 hours). The principal reason to use eptifibatide for PCI is to prevent platelet aggregation and the associated ischemia and myocardial infarction (MI). With improved laminar flow following stenting, prolonged infusion of eptifibatide may no longer be necessary. We hypothesize that after successful stenting with good angiographic results, patients can have eptifibatide discontinued immediately without a higher risk of adverse ischemic outcome, i.e. death, MI or unplanned target vessel revascularization (TVR) by 30 days. MI is defined as creatine kinase-MB (CK-MB) concentrations elevated to more than three times the upper limit of normal or new pathologic Q wave as seen on electrocardiograms (ECG). In order to prove this hypothesis, we estimate a sample size of 2,100 patients.

Before embarking on a large-scale clinical trial, we propose a pilot study using serum troponin I elevation as a surrogate end-point. Troponin I is a sensitive biomarker of ischemic injury. The absence of troponin I release following PCI would suggest excellent short and intermediate term prognosis. For the pilot study, we seek to prove the hypothesis that following successful PCI with stenting, an abbreviated regimen of eptifibatide is not inferior to the standard infusion in preventing ischemic injury, defined as troponin I release if baseline value is normal, or as CK-MB more than 3 times upper limit of normal if baseline troponin I is elevated. For this pilot study, we estimate a sample size of 620 patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female subjects
* 18 years of age or older
* Received aspirin, clopidogrel, heparin (unfractionated or low molecular weight [LMW]) and eptifibatide
* Had a successful PCI procedure with at least one stent deployed
* Availability of a hospital bed

Exclusion Criteria:

* Use of alternative anti-thrombin therapy during PCI (e.g. bivalirudin)
* High risk patients:
* Acute ST elevation MI < 48 hours (either direct PCI or rescue PCI)
* Unprotected left main PCI
* Obvious large thrombus on angiography
* Use of rotablation, atherectomy, or thrombectomy devices
* Unsatisfactory PCI results:
* Final thrombolysis in myocardial infarction (TIMI) flow < 3
* High grade dissection (> type B, if not completely resolved at completion of PCI)
* Evident or suspected thrombus
* Distal embolization
* Suboptimal stenting (> 20% residual stenosis)
* Side branch closure (≥ 1.5 mm branch or with associated symptoms)
* Abrupt closure during procedure (if prolonged > 15 min or not resolved at completion of PCI)
* Clinical instability
* Prolonged ischemia during PCI (> 15 min)
* Increased hazard of eptifibatide infusion:
* Unsatisfactory deployment of a closure device (if used)
* Large peri-procedure hematoma making the continuation of eptifibatide hazardous
* Any condition that will increase the hazard of continuing eptifibatide
* Operator discretion
* No informed consent
* Active participation in other research studies (unless with special exemption)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 624 (Actual)
Dates: Start 2004-12; Primary Completion 2007-07 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Ischemic injury is defined as troponin I release by 24 hours when the baseline troponin I is normal or by measuring creatine kinase (CK-MB) when the baseline troponin I is elevated. | 24 Hours

SECONDARY OUTCOMES:
30-day all-cause mortality, non-fatal myocardial infarction (MI), and unplanned target vessel revascularization (TVR) | 30 days
Composite event rate of non-coronary artery bypass graft (CABG) major bleeding, all-cause mortality, non-fatal MI, and urgent TVR at 30 days post PCI. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Fung, MB,BS, FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Saw J, Densem C, Walsh S, Jokhi P, Starovoytov A, Fox R, Wong G, Buller C, Ricci D, Mancini GB, Fung A. The effects of aspirin and clopidogrel response on myonecrosis after percutaneous coronary intervention: a BRIEF-PCI (Brief Infusion of Intravenous Eptifibatide Following Successful Percutaneous Coronary Intervention) trial substudy. JACC Cardiovasc Interv. 2008 Dec;1(6):654-9. doi: 10.1016/j.jcin.2008.08.017. PMID 19463380
- [Result] Fung AY, Saw J, Starovoytov A, Densem C, Jokhi P, Walsh SJ, Fox RS, Humphries KH, Aymong E, Ricci DR, Webb JG, Hamburger JN, Carere RG, Buller CE. Abbreviated infusion of eptifibatide after successful coronary intervention The BRIEF-PCI (Brief Infusion of Eptifibatide Following Percutaneous Coronary Intervention) randomized trial. J Am Coll Cardiol. 2009 Mar 10;53(10):837-45. doi: 10.1016/j.jacc.2008.09.060. PMID 19264239